CLINICAL TRIAL: NCT04346004
Title: Effect of Preoperative Iron Isomaltoside 1000 Administration on Hemoglobin Concentration in Patients Undergoing Transcatheter Aortic Valve Implantation: a Randomized Clinical Trial
Brief Title: Effect of Preoperative Iron Isomaltoside 1000 Administration on Hemoglobin Concentration in Patients Undergoing Transcatheter Aortic Valve Implantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2020-0143
Record Dates: First submitted 2020-04-06; First posted 2020-04-15 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Aortic Stenosis (Treated With TAVI)
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Saline Solution; iron isomaltoside 1000

STUDY DESIGN:
Intervention Model Description: Patients are divided into 2 groups, who are administered Iron isomaltoside & Vitamin B12 or who are administered Normal saline (N/S).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither participants, all care providers, investigators nor outcomes assessors know the treatment allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Participants in this group are administered N/S.
  Interventions: Drug: Normal saline
- Iron isomaltoside group (Experimental): Participants in this group are administered Iron isomaltoside & Vitamin B12.
  Interventions: Drug: Iron isomaltoside

INTERVENTIONS:
Drug: Normal saline — Participants in "Control group" are administered IV 100cc normal saline & IM normal saline (1cc) 1 day before surgery.
  Arms: Control group
Drug: Iron isomaltoside — Participants in "Iron isomaltoside group" are administered IV Iron maltoside diluted in 100 cc normal saline (20mg/kg, maximum dose: 1g) & IM Vitamin B12 (1mg) 1 day before surgery.
  Arms: Iron isomaltoside group

SUMMARY:
Transcatheter aortic valve implantation (TAVI) is a standard procedure for severe aortic stenosis patients with moderate or higher risk of surgery. Several studies have reported the adverse effects of blood disorders, such as anemia and iron deficiency, on the prognosis of patients undergoing TAVI, and many other studies have been conducted to find ways to prevent them.

Iron isomaltoside, the latest intravenous iron supplement, can effectively replenish iron store with a single high-dose injection. Research has shown that a preoperative single high-dose iron isomaltoside (1000mg) safely increased hemoglobin levels after surgery in patients undergoing cardiac surgery. However, there have been no studies on the effect of ultra-short-term use of intravenous iron supplements prior to TAVI procedure.

Therefore, we investigate the effect of a single high-dose of iron isomaltoside (20mg/kg, maximum dose: 1g) on the hemoglobin concentration after the TAVI.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 60 years and undergoing transcatheter aortic valve implantation (TAVI)

Exclusion Criteria:

* Emergency operation
* Cardiogenic shock or ventricular-assist device (eg. ECMO, IABP)
* Infectious condition
* Active bleeding
* Hypokalemia
* Severe chronic kidney disease (GFR(CKD-EPI) <30mL/min/1.73m2) or Dialysis
* Patients taking erythropoietin
* Aplastic anemia, Hemolytic anemia
* Hemochromatosis, Hemosiderosis
* Uncompensated liver cirrhosis, Acute hepatitis, Alcoholism
* Peptic / Duodenal ulcer, Crohn's disease, Ulcerative colitis
* Allergy to iron supplements or vitamin B12
* Symptomatic asthma, eczema
* Immunologic disease (e.g. Rheumatoid arthritis, Systemic lupus erythematosus)
* Malignancy
* Patients being treated in the intensive care unit due to heart failure or other major complications
* Patients who participated in other clinical studies that could affect prognosis
* Patients who cannot understand the informed consent (eg. Foreigner)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin (Hb) concentration | 1~3 days before TAVI (Baseline)
  Compare the Hb concentrations between the Iron isomaltoside group and the Control group.
Hemoglobin (Hb) concentration | within 5 minutes after TAVI
  Compare the Hb concentrations between the Iron isomaltoside group and the Control group.
Hemoglobin (Hb) concentration | 2 days after TAVI
  Compare the Hb concentrations between the Iron isomaltoside group and the Control group.
Hemoglobin (Hb) concentration | 2 weeks after TAVI (when the participant has not been discharged for 2 weeks) or 1st outpatient visit after TAVI (when the participant has been discharged within 2 weeks)
  Compare the Hb concentrations between the Iron isomaltoside group and the Control group.

SECONDARY OUTCOMES:
Transfusion requirement | 1~3 days before TAVI (Baseline)
  Compare the transfusion requirement between the Iron isomaltoside group and the Control group.
Transfusion requirement | During hospitalization period after TAVI, an average of 1 week
  Compare the transfusion requirement between the Iron isomaltoside group and the Control group.
Transfusion requirement | During 2 weeks after TAVI (when the participant has not been discharged for 2 weeks) or until 1st outpatient visit after TAVI (when the participant has been discharged within 2 weeks)
  Compare the transfusion requirement between the Iron isomaltoside group and the Control group.
Functional performance - Essential frailty toolset (EFT) | 1~3 days before TAVI (Baseline)
  Compare the functional performance between the Iron isomaltoside group and the Control group.
Functional performance - Handgrip | 1~3 days before TAVI (Baseline)
  Compare the functional performance between the Iron isomaltoside group and the Control group.
Functional performance - Essential frailty toolset (EFT) | 2 weeks after TAVI (when the participant has not been discharged for 2 weeks) or 1st outpatient visit after TAVI (when the participant has been discharged within 2 weeks)
  Compare the functional performance between the Iron isomaltoside group and the Control group.
Functional performance - Handgrip | 2 weeks after TAVI (when the participant has not been discharged for 2 weeks) or 1st outpatient visit after TAVI (when the participant has been discharged within 2 weeks)
  Compare the functional performance between the Iron isomaltoside group and the Control group.
Cognitive function - MMSE-K (Mini Mental State Exam) | 1~3 days before TAVI (Baseline)
  Compare the cognitive function between the Iron isomaltoside group and the Control group.
Cognitive function - MMSE-K (Mini Mental State Exam) | 2 weeks after TAVI (when the participant has not been discharged for 2 weeks) or 1st outpatient visit after TAVI (when the participant has been discharged within 2 weeks)
  Compare the cognitive function between the Iron isomaltoside group and the Control group.
Depression - SGDS-K (Short geriatric Depression Scale) | 1~3 days before TAVI (Baseline)
  Compare the depression between the Iron isomaltoside group and the Control group.
Depression - SGDS-K (Short geriatric Depression Scale) | 2 weeks after TAVI (when the participant has not been discharged for 2 weeks) or 1st outpatient visit after TAVI (when the participant has been discharged within 2 weeks)
  Compare the depression between the Iron isomaltoside group and the Control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine Anesthesia and Pain Research Institute Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No